CLINICAL TRIAL: NCT04274569
Title: Are Calcium- and Phosphate-containing Fluoride Varnishes More Effective Than Conventional Fluoride Varnish in Preventing Early Childhood Caries? A Randomized Clinical Trial.
Brief Title: Effect of Three Types of Fluoride Varnish in Preventing Early Childhood Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cynthia Kar-Yung Yiu, Clinical Professor in Paediatric Dentistry, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GRF Project HKU17106318
Record Dates: First submitted 2019-11-12; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Early Childhood Caries
Keywords: Caries; Fluoride vanish; Calcium phosphate; Randomised clinical trial; Remineralisation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium fluoride (NaF) (Active Comparator): Group 1: Quarterly application of a 5% NaF varnish (Duraphat® Varnish, Colgate-Palmolive Ltd, (UK) Ltd., Guildford, Surrey, UK)
  Interventions: Other: NaF vanish
- NaF plus tricalcium phosphate (TCP ) (Experimental): Group 2: Quarterly application of 5% NaF-TCP (ClinproTM White Varnish; 3M ESPE, St Paul, MN, USA)
  Interventions: Other: NaF-TCP
- NaF plus CPP-ACP (Experimental): Group 3: Quarterly application of a 5% NaF plus casein phosphopeptide-stabilized amorphous calcium phosphate complexes (CPP-ACP) (MI Varnish TM; GC corporation, Itabashi-Ku, Tokyo, Japan)
  Interventions: Other: NaF-CPP-ACP

INTERVENTIONS:
Other: NaF vanish — A disposable micro-brush will be used to apply the varnishes to all tooth surfaces. The fluoride varnish will be applied every 3 months, from baseline to 24-months follow-up.
  Arms: Sodium fluoride (NaF)
Other: NaF-TCP — A disposable micro-brush will be used to apply the varnishes to all tooth surfaces. The fluoride varnish will be applied every 3 months, from baseline to 24-months follow-up.
  Arms: NaF plus tricalcium phosphate (TCP )
Other: NaF-CPP-ACP — A disposable micro-brush will be used to apply the varnishes to all tooth surfaces. The fluoride varnish will be applied every 3 months, from baseline to 24-months follow-up.
  Arms: NaF plus CPP-ACP

SUMMARY:
This study evaluates and compares the effect of two types of calcium- and phosphate-containing fluoride varnishes to conventional fluoride varnishes in preventing early childhood caries.

DETAILED DESCRIPTION:
Fluoride vanish is the most commonly used professionally applied topical agent. Traditional fluoride vanish application has been reported to exhibit significant caries inhibiting effect in both permanent teeth and primary teeth. The greatest advantage of fluoride vanish is its ability to adhere to tooth tissues for a longer period of time that enables improved fluoride uptake. It allows continuous release of fluoride ions into enamel, dentine, plaque, and saliva.The main action of topical fluoride is to retard demineralization and promote remineralization of enamel by the uptake of calcium and phosphates from saliva. The proposed mechanism of action of topical fluoride is the formation of intraoral calcium fluoride reservoirs, which are retained on enamel and slowly released to inhibit mineral loss during demineralization.

However, the formation of the intraoral calcium fluoride reservoirs is limited by the availability of intraoral calcium and fluoride ions. Low concentration of salivary calcium and phosphate ions leads to mineral deposition only at the surface of enamel as a result of low ion concentration gradient. Deposition of minerals at the surface of enamel alone may not improve the structural properties of the deep part of the incipient carious lesions. Hence, many manufacturers have modified fluoride vanish to include calcium and phosphate ions in an attempt to further improve efficacy of fluoride varnishes.

The in vitro remineralizing effects of calcium- and phosphate-containing fluoride vanishes are encouraging and scientifically sound, a longitudinal, high quality clinical study is needed to verify the laboratory findings.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy children age between 3-4 of age with unremarkable medical history and at high caries risk with at least one carious lesion (precavitated or cavitated) (Agouropoulos et al 2014). The high caries risk children are chosen because it is anticipated that they will benefit more from the topical fluoride varnish application than the low caries risk children.

Exclusion Criteria:

* Patients who had received professional fluoride application in the past 6 months

  * Patients with underlying medical history or special health care needs
  * Patient who are uncooperative or refuse the treatment
  * Patient who are allergic to milk protein (as MI VarnishTM contains "casein, a milk protein)
  * Patient with contraindication for fluoride varnish e.g. hypersensitivity to colophony and/or any other constituents
  * Patient who have primary teeth with enamel hypoplasia

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 570 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with new caries and new dmfs. | 24 months

SECONDARY OUTCOMES:
MS growth | 12 months and 24 months
  Quantity of mutans streptococcus (MS) measured by quantitative polymerase chain reaction (qPCR)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No